CLINICAL TRIAL: NCT01715389
Title: Evaluation of a Shared Decision Making Portal for Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-009407
Record Dates: First submitted 2012-10-10; First posted 2012-10-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Asthma
Keywords: Asthma; Goals; Shared Decision Making; Patient Portal; Electronic Medical Record
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Parents in the intervention group will use the MyAsthma Patient Portal to receive enhanced educational information on asthma and its treatment, identify concerns and goals related to asthma treatment, track progress toward goals and management of concerns monthly, and track asthma symptoms monthly.
  Clinicians seeing intervention families at office visits will have access to information from the portal including concerns, goals, progress toward goals, and tracking of asthma symptoms.
  Interventions: Other: MyAsthma Patient Portal
- Control (No Intervention): The control group will be signed up for MyChart but not use the MyAsthma Patient Portal. This group will be referred to asthma educational content on the CHOP website, complete study measures and otherwise, receive standard care.

INTERVENTIONS:
Other: MyAsthma Patient Portal — Parents in the intervention group will use the MyAsthma Patient Portal to receive enhanced educational information on asthma and its treatment, identify concerns and goals related to asthma treatment, track progress toward goals and management of concerns monthly, and track asthma symptoms monthly.
  Clinicians seeing intervention families at office visits will have access to information from the portal including concerns, goals, progress toward goals, and tracking of asthma symptoms.
  Arms: Intervention

SUMMARY:
This pilot intervention study will test the feasibility and acceptability and explore the outcomes of a primary care-based shared decision making (SDM) electronic medical record (EMR)-based portal that provides education, elicits and tracks patients/families' treatment concerns and goals, assesses symptoms and asthma control over time, and provides decision support to clinicians and families.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians of children aged 6-12 with persistent asthma, currently receiving chronic maintenance therapy, cared for at a study practice, with consistent access to a computer with an internet connection where they feel comfortable accessing MyChart (patient portal)
* Clinician at study site

Exclusion Criteria:

* parents non-english speaking
* child's primary care provider at the time of enrollment is a pediatric resident
* not meeting inclusion criteria

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention to parents and clinicians | 24 months
  Parents and clinicians will be asked a series of open-ended questions regarding themes including satisfaction, acceptability and unintended consequences of using the portal for intervention subjects and using MyChart in general for control subjects. Subjects will also be asked a series of Likert-scaled questions related to satisfaction.

SECONDARY OUTCOMES:
Shared decision making | Baseline
  Joint participation in decision-making will be measured by the Observing Parent Involvement (OPTION) scale.
Parent Activation | 0 months, 3 months, 6 months
  Parent activation will be measured by the Parent Patient Activation Measure (PPAM).
Goal Attainment | 0 months, 3 months, 6 months then Monthly
  Parents will identify one or more goals at the study start. Progress toward the goal(s) will be assessed at 3 and 6 month follow-up using Likert-scaled items for the control group, and monthly through use of the portal for the intervention group.
Asthma-Related Quality of Life | 0 months, 6 months
  Asthma-related quality of life will be measured using The Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF)
Asthma Control | 0 months, 6 months
  Asthma control will be assessed using the Pediatric Asthma Control Tool (PACT)
Asthma-related Utilization | 3 months, 6 months
  Utilization will be measured by parent report and chart review by the research team of the following:
  Any primary care or subspecialty outpatient encounters relevant to asthma care, asthma-specific acute primary care visits or Urgent Care Center visits, asthma-specific Emergency Room visits, asthma-specific hospital admissions.
Asthma Medication Adherence/Receipt | 6 months
  Prescribed medications for the treatment and management of asthma Type and number of prescriptions for asthma
Feasibility of Recruitment | 24 months
  The feasibility of recruitment will be assessed by examining the proportion of all families contacted who meet enrollment criteria and the proportion of families meeting enrollment criteria who enroll.
Feasibility of Follow-up | 24 months
  The feasibility of follow-up will be assessed by the proportion of enrolled families who complete each study measure.
Feasibility of Portal Use | 24 months
  The feasibility of portal use will be assessed by the level of research team/other outside support needed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Fiks, MD, MSCF, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States